CLINICAL TRIAL: NCT00607945
Title: Dietary Fatty Acids As Complementary Therapy in Type 2 Diabetes Mellitus
Acronym: FACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); GlaxoSmithKline (Industry); Bunge Loders Croklaan (Industry); LifeScan (Industry)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007H0185; R21AT003520-01A2 (NIH); 5R21AT003520 (NIH)
Record Dates: First submitted 2008-01-24; First posted 2008-02-06 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; conjugated linoleic acid; weight loss; rosiglitazone; glucose control; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss; Insulin Resistance | interventions — Rosiglitazone; Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0 g CLA (Placebo Comparator): Avandia (Rosiglitazone) 4-8mg/day OR other diabetes medication currently prescribed to participant, 0 g CLA, 8 g Placebo oil (based on typical American diet)
  Interventions: Drug: Rosiglitazone (Avandia) OR other diabetes medication currently prescribed to participant
- 3.2 g CLA (Experimental): Avandia 4-8mg/day OR other diabetes medication currently prescribed to participant, 3.2 g CLA, 4.8 g placebo oil (based on typical American diet)
  Interventions: Drug: Rosiglitazone (Avandia) OR other diabetes medication currently prescribed to participant; Dietary Supplement: conjugated linoleic acid (CLA)
- 6.4 g CLA (Experimental): Avandia 4-8mg/day OR other diabetes medication currently prescribed to participant, 6.4 g CLA, 1.6 g placebo oil (based on typical American diet)
  Interventions: Drug: Rosiglitazone (Avandia) OR other diabetes medication currently prescribed to participant; Dietary Supplement: conjugated linoleic acid (CLA)

INTERVENTIONS:
Drug: Rosiglitazone (Avandia) OR other diabetes medication currently prescribed to participant — Rosiglitazone 4-8mg/day, pill, from week -4 to week 32 OR other diabetes medication taken as prescribed from week -4 to week 32
  Other Names: Avandia
Dietary Supplement: conjugated linoleic acid (CLA) — 3.2 g/day, capsule, week 0 to week 32
  Other Names: Tonalin, Clarinol
  Arms: 3.2 g CLA
Dietary Supplement: conjugated linoleic acid (CLA) — 6.4 g/day, capsule, week 0 to week 32
  Other Names: Tonalin, Clarinol
  Arms: 6.4 g CLA

SUMMARY:
The purpose of the study is to see how a dietary oil called conjugated linoleic acid, or CLA, might be useful in combination with diabetes medication. Some studies show that CLA can modestly reduce body weight and body fat. Our research idea is that taking CLA will reduce body weight and body fat without interfering with the diabetes medications' effects on blood sugar.

DETAILED DESCRIPTION:
The long term goal of this research is to develop effective complementary strategies to aid in the management of type 2 diabetes (T2DM). Our central hypothesis is that CLA reduces body weight and body fat mass when administered concomitantly with oral diabetes medication, The rationale of this study is that using CLA to reduce body weight and body fat in people with T2DM may improve efficacy and longevity of the oral diabetes medications in the management of T2DM. We plan to test our central hypothesis and accomplish the overall objective of this research by pursuing the following three specific aims.

Specific Aim 1: Determine the ability of CLA to reduce body weight and body fat mass in people using oral diabetes medication for management of T2DM.

Specific Aim 2: Determine the ability of CLA to modulate insulin sensitivity when combined with oral diabetes medication.

Specific Aim 3: Determine the safety and tolerability of CLA in combination with oral diabetes medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* HbA1c ≤ 9%
* Overweight or obese (BMI ≥ 25 kg/m2 and ≤ 45 kg/m2)
* Age ≥ 30 and ≤ 70 years (postmenopausal if female)
* Stable medical therapy for past 3 months
* Stable body weight (within ± 2 kg) for past 3 months
* Plans to remain in the Columbus, OH metropolitan area for at least 1 year

Exclusion Criteria:

* Substance abuse
* Current use of prescription or over-the-counter medications or supplements known to affect body composition
* Current use of prescription or over-the-counter medications or supplements known to interact with thiazolidinediones(TZDs)
* Current or previous diagnosis of congestive heart failure
* Self-report of claustrophobia
* Abnormal liver function
* Impaired cognitive function
* Current or previous diagnosis of renal disease
* Gastrointestinal diseases or disorders
* Current use of hormone therapies, or use within the past 3 months
* Discontinuation of diabetes medication

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference in change in body weight of the intervention groups | Between baseline and week 32, or end of study

SECONDARY OUTCOMES:
Change in fat mass | Between baseline and week 32
Change in lean mass | Between baseline and week 32
Change in insulin sensitivity | Between week 0 and week 32
Change in lipid profile (TChol, LDL, HDL, C-reactive protein) | Weeks -4, -1, 0, 8, 16, 24, 31, 32
Changes in adipocytokine profile (leptin, adiponectin, visfatin, and resistin) | Weeks -4, -1, 0, 8, 16, 24, 31, 32
Changes in liver enzymes (ALT and AST) | Weeks -4, -1, 0, 8, 16, 24, 31, 32
Edema | Weeks -4, -1, 0, 8, 16, 24, 31, 32
Change in glucose control | Weeks -1, 16, 31
Change in bone density, bone formation and resorption markers | Weeks -4, -1, 31
Change in C-Peptide | Weeks - 4, -1, 0, 1, 8, 16, 24, 31, 32
Diabetes coping behaviors and self-efficacy | Weeks -4, -1, 32
Chronic stress (as measured by questionnaire) | Weeks -4 and 32
Appetite (as measured by appetite rating scale) | Weeks -4, 0, 16, 32
EKG | Weeks -4, 16, 32
BNP (brain type natriuretic peptide) | Weeks -4 and 32
Energy balance (physical activity recalls, food records, indirect calorimetry) | Weeks -1, 16, 31
Compliance (fatty acid composition, pill counts) | Weeks -1, 0, 8, 16, 24, 31, 32
Nutrition knowledge | Weeks -4, 0, 32

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Belury, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Clinical Research Center (Davis Medical Research Center), Columbus, Ohio, United States